CLINICAL TRIAL: NCT05390229
Title: Comparison of the Performance of Diagnostic Contrast-enhanced Mammography and Magnetic Resonance Imaging for Suspicious Breast Lesion At Screening
Brief Title: Screening Contrast-enhanced Mammography
Status: Recruiting | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-4432
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of this study is to compare the diagnostic performance of two diagnostic methods, namely CESM and MRI, in the evaluation of a lesion suspicious of breast cancer in 300 Quebec women referred for the investigation of breast cancer. breast lesion suspected of cancer. All suspicious lesions will be evaluated by these two diagnostic imaging and by TNM. Then, radiologists will respectively interpret diagnostic imaging, without knowing the result of the other imaging in parallel with the study. The sensitivity, specificity, positive predictive value and negative predictive value for his diagnostic imaging will then be determined. Histopathological confirmation by biopsy or surgery will be used as a standard value.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 and over
* At least one breast lesion with BIRADS classification 5

Exclusion Criteria:

* Refusal to perform the biopsy or surgery
* Pregnant or possibly pregnant woman
* Usual contraindication to contrast product

  * Significant kidney failure
  * Allergy to contrast medium
* hyperthyroidism
* Usual contraindications to MRI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients referred to the breast clinic at the HSS for a mass suspected of cancer (BIRAD 5) will potentially be considered in the study. These women come either from the Quebec breast cancer screening program, or referred by their attending physician in the investigation of a palpable/symptomatic mass or in an investigation requested for a high-risk patient. These patients will then be referred to us by the attending surgeons as part of the preoperative evaluation of the lesion. Preoperatively, mammography (standard or by tomosynthesis) is considered standard and MRI can also be requested as standard by the surgeon. The patients included will be those for whom an MRI will be prescribed. All patients will receive diagnostic imaging (CESM, MRI and TMN) within 30 days of surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value for breast cancer | Breast cancer screening
  To measure sensitivity, specificity, positive predictive value and negative predictive value for CESM and MRI using histopathological confirmation as a standard value.
Diagnostic value for suspicious breast lesion | Breast cancer screening
  To determine the ability of diagnostic imaging to identify other breast masses suspicious of cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- St-Sacrement Hospital, Québec, Quebec, Canada